CLINICAL TRIAL: NCT06600802
Title: Intrinsic Validity of Molecular Marker(s) Detection on Tissular Tumoral DNA to Predict the Efficacy of 177Lutetium-PSMA-617 (Lu-PSMA) Treatment for Castration-resistant Metastatic Prostate Cancer (PSMA-PRED)
Brief Title: Intrinsic Validity of Molecular Marker(s) Detection on Tissular Tumoral DNA to Predict the Efficacy of 177Lutetium-PSMA-617 (Lu-PSMA) Treatment for Castration-resistant Metastatic Prostate Cancer
Acronym: PSMA-PRED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Jean Perrin (Other)
Collaborators: GIRCI Auvergne Rhône-Alpes (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-A00246-41
Record Dates: First submitted 2024-07-22; First posted 2024-09-19 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Castration-resistant Metastatic Prostate Cancer; Treated by 177Lutetium-PSMA-617 (Lu-PSMA)
Keywords: mCRPC; Lu-PSMA; biomarkers; response; prediction
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): Genetic analysis will be conducted on intial tumor sample in order to identify biomarkers
  Interventions: Biological: Blood samples

INTERVENTIONS:
Biological: Blood samples — A total of 3 blood samples (2 tubes of 9mL each) are added. The first sample will be taken at the inclusion visit, the 2nd at the end of the 2nd treatment cycle and the last at the end of Lu-PSMA treatment.

SUMMARY:
Prostate cancer is the most common cancer in men. Its incidence is rising as the population ages. In the localized stage, the 5-year overall survival rate (OS) is 98%. Metastatic progression and resistance to castration have a negative impact on prognosis. Despite recent advances in management, the 5-year OS is around 30%. Therapeutic advances in this indication have been made mainly by the use of taxanes and second-generation hormone therapy. These treatments have improved OS and progression-free survival (PFS). They are now used as standard therapy.

More recently, the Phase III VISION trial confirmed the improvement in OS and radiological PFS achieved by treatment with the radioligand 177Lutetium-PSMA-617 (Lu-PSMA) in patients with advanced metastatic castration-resistant prostate cancer (mCRPC).

This treatment is currently available in early access in France. Despite encouraging results, 40% of patients will not respond to Lu-PSMA, and there are currently no validated predictive factors. Studies are currently on going, but the identification of biomarkers seems necessary to better stratify risk in these patients.

Numerous tissue prognostic tests based on molecular characteristics or cell proliferation are emerging with this in mind. At present, molecular profiling is not a routine technique for prostate cancer, as it is for other solid cancers. At an early stage, the Decipher® Genomic classification tool has shown prognostic utility independently of therapeutic and clinico-pathological data.

According to recent studies, methylome analysis would enable the subdivision of mCRPCs and could help identify new therapeutic targets.

In the metastatic phase, certain molecular abnormalities involving DNA repair genes are predictive of response to PARP inhibitors.

Molecular analysis (mutations, copy number alterations, gene expression, DNA methylation) could therefore be useful in optimizing the management of mCRPC patients treated with Lu-PSMA.

If reliable molecular abnormalities are identified on tissue, a diagnostic technique based on circulating tumor DNA (ctDNA) analysis will be useful in decision-making for these patients. A biological collection will therefore be created during the course of this study, with a view to using ctDNA analysis in subsequent research.

DETAILED DESCRIPTION:
Prostate cancer is the most common cancer in men. Its incidence is rising as the population ages. In the localized stage, the 5-year overall survival rate (OS) is 98%. Metastatic progression and resistance to castration have a negative impact on prognosis. Despite recent advances in management, the 5-year OS is around 30%. Therapeutic advances in this indication have been made mainly by the use of taxanes and second-generation hormone therapy. These treatments have improved OS and progression-free survival (PFS). They are now used as standard therapy.

More recently, the Phase III VISION trial confirmed the improvement in OS and radiological PFS achieved by treatment with the radioligand 177Lutetium-PSMA-617 (Lu-PSMA) in patients with advanced metastatic castration-resistant prostate cancer (mCRPC).

This treatment is currently available in early access in France. Despite encouraging results, 40% of patients will not respond to Lu-PSMA, and there are currently no validated predictive factors. Studies are currently on going, but the identification of biomarkers seems necessary to better stratify risk in these patients.

Numerous tissue prognostic tests based on molecular characteristics or cell proliferation are emerging with this in mind. At present, molecular profiling is not a routine technique for prostate cancer, as it is for other solid cancers. At an early stage, the Decipher® Genomic classification tool has shown prognostic utility independently of therapeutic and clinico-pathological data.

According to recent studies, methylome analysis would enable the subdivision of mCRPCs and could help identify new therapeutic targets.

In the metastatic phase, certain molecular abnormalities involving DNA repair genes are predictive of response to PARP inhibitors.

Molecular analysis (mutations, copy number alterations, gene expression, DNA methylation) could therefore be useful in optimizing the management of mCRPC patients treated with Lu-PSMA.

If reliable molecular abnormalities are identified on tissue, a diagnostic technique based on circulating tumor DNA (ctDNA) analysis will be useful in decision-making for these patients. A biological collection will therefore be created during the course of this study, with a view to using ctDNA analysis in subsequent research.

This is an interventional, multi-center study. The study is prospective, single-arm, open-label and non-randomized.

Its primary objective is to identify biomarkers of interest, in primary tissue, predictive of response to Lu-PSMA treatment in patients with mCRPC, through the detection of molecular abnormalities in DNA/RNA and methyloma.

ELIGIBILITY:
Inclusion Criteria:

* Male >18 years of age
* ECOG ≤ 2
* Patient with histologically confirmed of metastatic castration resistant prostatic adenocarcinoma and with tumor biological material available (prostatic biopsies or prostatectomy)
* Patient who received at least one taxane line and a second generation hormone therapy line
* Patient receiving androgen deprivation therapy with serum testosterone < 50 ng/dL or < 1.7 nmol/L or having undergone surgical castration
* Progressive mCRPC based based on at least 1 of the following criteria :

  * Serum or plasma PSA progression defined as 2 consecutive increases in PSA measured at least 1 week prior. The minimal start value is 2.0 ng/mL ; 1,0 ng/mL is the minimal start value if confirmed increase in PSA is the only indication of progress
  * Soft-tissue progression by RECIST 1.1 criteria
  * Progression of bone disease : two new lesions ; only the positivity of bone scan defines metastatic bone disease, according to PCWG3 criteria.
* Patients with at least one metastasis, bone and/or soft tissue and/or visceral, documented by the following methods in the 43 days prior to inclusion :

  * Bone metastasis (regardless of location) highlighted by bone scan AND/OR
  * Lymph nodes metastasis, regardless of size and location; if the metastasis are only lymph nodes, the short axis of at least one node should be at least 15 mm AND outside the pelvis ; AND/OR
  * Visceral metastasis, regardless of size and location; a history of visceral metastasis at any time prior to randomization should be encoded as the presence of visceral metastasis at baseline (i.e., a patient with visceral metastasis prior ADT introduction which are disappeared at baseline will be counted as having visceral metastasis and will be considered to have a high tumor volume during stratification)
* Patient with Lu-PSMA treatment indication, confirmed by PET 68Ga-PSMA-11. Eligibility for 68Ga-PSMA-11 PET is defined as:

  * At least one lesion with a binding intensity greater than that of the liver parenchyma (definition of positivity),
  * All lymph node lesions larger than 25 mm in the short axis must be positive on PSMA PET
  * All bone metastases with a soft tissue component ≥ 10 mm in the largest diameter must be positive on PSMA-PET
  * All solid organ metastases (e.g., lung, liver, adrenal glands, etc.) ≥ 10 mm in the largest diameter must be positive on PSMA-PET.
* Adequate organ function :

  * Bone marrow reserve :

    * Absolute neutrophil count ≥ 1.5 x 10^9/L
    * Platelets ≥ 100 x 10^9/L.
    * Hemoglobin ≥ 9 g/dL
  * Hepatic function :

    * Total bilirubin ≤ 2 x the upper limit of normal (ULN). For participants with known Gilbert's Syndrome ≤ 3 x ULN is permitted.
    * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3.0 x ULN OR ≤ 5.0 x ULN for patients with liver metastases.
    * Albumin > 2.5 g/dL
  * Renal function : Glomerular Filtration Rate (GFR) ≥ 50 mL/min/1.73m2 according to MDRD equation.
* Obtaining the patient's free and informed consent
* Social security scheme or beneficiary.

Exclusion Criteria :

* Continuation of second-generation hormone therapy Patient
* Other cancer in the last 3 years likely to change life expectancy or interfere with the assessment of the disease
* Protected adult
* History of somatic or psychiatric illness/condition that may interfere with study objectives and evaluations
* Patient unable to understand and comply with study instructions and requirements
* ECOG > 2
* Dilation of pyelocalicial cavities not previously supported
* Obstruction of bladder discharge or uncontrollable and simultaneous urinary incontinence
* Symptomatic spinal cord compression or clinical or radiological findings indicating imminent spinal cord compression
* Fractured risk of bone damage
* Active and symptomatic brain injury
* Concurrent participation in a therapeutic trial and administration of any investigational agent within 28 days of inclusion
* Metastatic tumor tissue as the only material available for prostate cancer diagnosis
* Previous treatment with any of the following in the 6 months prior to inclusion : Strontium-89, Samarium-153, Rhenium-186, Rhenium-188, Radium-223, hemi-cyclic irradiation
* Previous treatment with radioligands targeting PSMA
* Known hypersensitivity to one of the study treatments or its excipients or similar class drugs
* Transfusion or use of bone marrow stimulating agents for the sole purpose of making a participant eligible for inclusion in the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2034-06-30 (Estimated); Study Completion 2034-06-30 (Estimated)

PRIMARY OUTCOMES:
Molecular abnormalities retained on primary tumor sample predicting response to Lu-PSMA in metastatic castration resistant prostate cancer patients assessed according to RECIST 1.1 and/or PCWG3 criteria | From enrollment to 24 months after Lu-PSMA treatment
  Biological interpretation and response to Lu-PSMA treatment on bone scan and CT scan according to RECIST 1.1 and/or PCWG3 criteria

SECONDARY OUTCOMES:
Correlation between biomarker(s) (molecular abnormalities retained on primary tumor sample for the first outcome measure) and survival without radiological progression | From enrollment to 24 months after Lu-PSMA treatment
  Radiological progression free survival defined as the duration between the start date of treatment and the date of the first progression of the disease according to criteria RECIST V1.1 and criteria PCWG3; or the date of death whatever the cause.
Correlation between biomarker(s) (molecular abnormalities retained on primary tumor sample for the first outcome measure) and survival without biological progression | From enrollment to 24 months after Lu-PSMA treatment
  Biological progression free survival defined as the duration between the start date of treatment and the date of the first PSA progression
Correlation between biomarker(s) (molecular abnormalities retained on primary tumor sample for the first outcome measure) and survival without clinical progression | From enrollment to 24 months after Lu-PSMA treatment
  Clinical progression free survival, definieds as the duration between the treatment start date and the date of the first clinical progression
Correlation between biomarker(s) (molecular abnormalities retained on primary tumor sample for the first outcome measure) and overall survival | From enrollement to the end of the study, up to 58 months
  Overall survival definied as the time interval between the start date of treatment and the date of death whatever the cause
Correlation between the biomarker(s) (molecular abnormalities retained on primary tumor sample for the first outcome measure) and adverse effects during treatment. | From enrollment to the end of Lu-PSMA treatment, up to 58 months
  Toxicities related to treatment of grade 3 or higher according to CTCAE v. 5.0 and any EIG
Assess whether consideration of clinical characteristics improves biomarker performance | From enrollement to end of Lu-PSMA treatment, up to 58 months
  Performance status (0 to 4), pain and adverse events evaluations as assessed by CTCAE v4.0
Assess whether consideration of radiological characteristics improves biomarker performance | From enrollement to end of Lu-PSMA treatment, up to 58 months
  Radiological evaluation as assessed by RECIST criteria V1.1 and PCWG3 criteria
Assess whether consideration of biological characteristics improves biomarker performance | From enrollement to end of Lu-PSMA treatment, up to 58 months
  Biological evaluation as assessed with PSA level
Biological interpretation and response to Lu-PSMA treatment on PET scan | From enrollment to 24 months after Lu-PSMA treatment
  Radiological progression free survival defined as the duration between the start date of treatment according to RECIP 1.0 criteria for patients who underwent 68Ga-PSMA-11 PET scans

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Centre Jean PERRIN, Clermont-Ferrand
  - CHU de Grenoble, La Tronche
  - Hospices Civiles de Lyon, Pierre-Bénite
  - Hôpital privé de la Loire, Saint-Etienne
  - Centre Paul STRAUSS, Strasbourg